CLINICAL TRIAL: NCT05994859
Title: Y-90 Selective Internal Radiation Therapy for Potentially Resectable Hepatocellular Carcinoma: a Prospective, Single Arm Trial
Brief Title: SIRT for Potentially Resectable HCC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIIR-15
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; unresectable; selective internal radiation therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sirtuins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SIRT (Experimental): Treatment with SIRT.
  Interventions: Procedure: SIRT

INTERVENTIONS:
Procedure: SIRT — The patients will receive 1-2 sessions of SIRT. If the patients have invasive tumors, extensive liver involvement or vascular invasion, systematic treatment will be added.

SUMMARY:
This study is conducted to evaluate the efficacy and safety of Y-90 selective internal radiation therapy (SIRT) in patients with potentially resectable hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
This is a bi-center, prospective study to evaluate the efficacy and safety of SIRT in patient with potentially resectable HCC.

35 patients with potentially resectable (initially unresectable) HCC will be enrolled in this study. The patients will receive 1-2 sessions of SIRT. If the patients have invasive tumors, extensive liver involvement or vascular invasion, systematic treatment will be added. If the patients are evaluated as resectable during follw-up, liver resection will be recommended.

The primary end point of this study is success rate of conversion to resection. The secondary endpoints are objective response rate (ORR), disease control rate (DCR), progression-free survival (PFS), time to progression (TTP), duration of response (DOR), overall survival (OS) and adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

* HCC with diagnosis confirmed pathologically or clinically
* No pervious treatment for HCC
* At least one measurable intrahepatic target lesion
* Potentially resectable HCC: tumor(s) confined to the left/right hemiliver, with/without invasion to the unilateral branch of the portal vein and/or hepatic vein
* Disease amenable to SIRT (after evaluation)
* Child-Pugh Class A or without cirrhosis
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1
* Patients with active hepatitis B are allowed, but they need to receive antiviral treatment to achieve a HBV DNA<10^3 IU/mL
* Patients with hepatitis C need to finish the anti-HCV treatment
* Adequate organ and bone marrow function; the blood biochemical examination: platelet count ≥75×10^9/L, white blood cell count >3.0×10^9/L, absolute value of neutrophils >1.5×10^9/L, hemoglobin ≥85 g/L, ASL and AST≤5×ULN, creatinine≤1.5×ULN, INR<1.5 or PT/APTT normal range
* Life expectancy of at least 6 months

Exclusion Criteria:

* Tumor involving main portal vein, bilateral branches of portal vein, or vena cava
* tumor extention beyond one lobe of the liver
* Bilobar tumor distribution
* Extrahepatic metastasis
* Decompensated liver function, including ascites, bleeding from esophageal and gastric varices, and/or hepatic encephalopathy
* Organ (heart, kidney) dysfunction
* HBsAg and anti-HCV antibody positive concurrently
* History of malignancy other than HCC
* Uncontrolled infection
* History of HIV
* History of organ and cell transplantation
* Patients with bleeding tendency

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2026-08-09 (Estimated); Study Completion 2027-02-09 (Estimated)

PRIMARY OUTCOMES:
Success rate of conversion to resection | 3 years
  The proportion of patients with initially unresectable HCC who were evaluated by the surgical team as suitable for second-stage surgical resection after SIRT

SECONDARY OUTCOMES:
Objective response rate (ORR) | 3 years
  The percentage of patients who have a best overall tumor response rating of complete response (CR) or partial response (PR)
Disease control rate (DCR) | 3 years
  The percentage of patients who have a tumor response rating of CR, PR, or stable disease (SD)
Progression-free survival (PFS) | 3 years
  The time between the first treatment and the first occurrence of disease progression (PD) or death from any cause, whichever occurs first
Time to progression (TTP) | 3 years
  the time interval from first treatment to the first occurrence of disease progression
Duration of response (DOR) | 3 years
  the time from initial objective response (CR or PR) until PD or death, whichever occurs first
Overall survival (OS) | 3 years
  The time from initiation of treatment until the date of death from any cause
Adverse Events (AEs) | 3 years
  Number of patients with AEs assessed by NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China